CLINICAL TRIAL: NCT04110535
Title: A Double-blind, Randomized Crossover Study to Assess the Subjective Abuse Potential of Intravenous Remimazolam Compared to Midazolam and Placebo in Recreational CNS Depressant Users
Brief Title: Abuse Potential of Intravenous Remimazolam Compared to Midazolam and Placebo in Recreational CNS Depressant Users
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Paion UK Ltd. (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CNS7056-014
Record Dates: First submitted 2019-09-27; First posted 2019-10-01 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Abuse, Drug
Keywords: remimazolam
MeSH Terms: conditions — Substance-Related Disorders | interventions — remimazolam; Midazolam; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Remimazolam 5 mg (Experimental): IV administration of remimazolam 5 mg
  Interventions: Drug: Remimazolam
- Remimazolam 10 mg (Experimental): IV administration of remimazolam 10 mg
  Interventions: Drug: Remimazolam
- Midazolam 2.5 mg (Active Comparator): IV administration of midazolam 2.5 mg
  Interventions: Drug: Midazolam
- Midazolam 5 mg (Active Comparator): IV administration of midazolam 5 mg
  Interventions: Drug: Midazolam
- Placebo (Placebo Comparator): Saline injection
  Interventions: Other: Saline

INTERVENTIONS:
Drug: Remimazolam — IV administration over 1 minute
  Other Names: CNS7056
  Arms: Remimazolam 10 mg; Remimazolam 5 mg
Drug: Midazolam — IV administration over 1 minute
  Arms: Midazolam 2.5 mg; Midazolam 5 mg
Other: Saline — IV administration over 1 minute
  Arms: Placebo

SUMMARY:
A double-blind, randomized crossover study to assess the subjective abuse potential of intravenous remimazolam compared to midazolam and placebo in recreational CNS depressant users

ELIGIBILITY:
Inclusion Criteria:

1. Must have provided written informed consent prior to the initiation of any protocolspecific procedures.
2. Male and female adults, between 18 and 55 years of age, inclusive.
3. Body mass index (BMI) within 19.0 to 33.0 kg/m2, inclusive (minimum weight of at least 50.0 kg at Screening).
4. Healthy, as determined by having no clinically significant medical history, physical examination, 12-lead ECG, vital signs, or laboratory (including hematology, clinical chemistry, urinalysis, and serology) findings, as judged by the investigator.
5. Recreational CNS depressant user, defined as follows:

   1. ≥ 10 lifetime non-therapeutic experiences (ie, for psychoactive effects) with CNS depressants (eg, benzodiazepines, barbiturates, opioids, zolpidem, zopiclone, propofol/fospropofol, gamma-hydroxybutyrate)
   2. ≥ 1 non-therapeutic use of a CNS depressant within the 8 weeks prior to Screening
   3. ≥ 1 non-therapeutic use of benzodiazepines within the 12 months prior to Screening
6. Must pass Qualification Phase (Drug Discrimination and Tolerability) eligibility criteria (Section 9.3.1 and 9.3.2, respectively).
7. Female subjects must be of non-childbearing potential (postmenopausal, with > 1 year since last menses and a follicular stimulating hormone (FSH) value > 40 mIU/mL, or surgically or congenitally sterile), or, if of childbearing potential, must be using and willing to continue using highly effective contraception, defined as methods of birth control that result in a low failure rate (ie, less than 1% per year) when used consistently and correctly, such as implants, injectables, combined oral contraceptives, some intrauterine devices, sexual abstinence, or a vasectomized partner, for at least 1 month prior to Screening (at least 3 months for oral and transdermal contraceptives) and for at least 14 days after last study drug administration.
8. Able to speak, read, and understand English sufficiently to allow completion of all study assessments.
9. Must be willing to comply with the requirements and restrictions of the study.

Exclusion Criteria:

1. Drug or alcohol dependence within the 12 months prior to Screening (except nicotine), as defined by the Diagnostic and Statistical Man ual of Mental Disorders, fourth edition, text revision (DSM-IV-TR), or any self-reported dependence or "addiction" within the subject's lifetime (except nicotine or caffeine).
2. Subjects who have ever been in treatment for substance use disorder(s) (except smoking cessation).
3. History or presence of any clinically significant cardiac, psychiatric, endocrine, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, renal, or other major disease at Screening, which in the opinion of the investigator would jeopardize the safety of the subject or the validity of the study results, including subjects with chronic renal failure or congestive heart failure.
4. In the opinion of the investigator, the subject was at risk for respiratory depression, including subjects with obstructive apnea, upper airway obstruction, chronic obstructive pulmonary disease, acute or severe bronchial asthma, hypercarbia, or other severe cardio-respiratory disease.
5. Positive for hepatitis B, hepatitis C, or human immunodeficiency virus (HIV).
6. History of, or evidence at the time for, suicidal ideation with intent, with or without a plan or method, in the past 5 years or suicidal behavior in their lifetime or those who were actively suicidal based on the Columbia-Suicide Severity Rating Scale (C-SSRS).
7. Unexplained significant and recent loss of consciousness, or history of significant head trauma with loss of consciousness.
8. Reported history of acute narrow-angle glaucoma.
9. Required concomitant treatment with any prescription or non-prescription medications (with the exception of hormonal contraceptives, hormone replacement, and acetaminophen) or natural health products (herbal remedies), including strong cytochrome P450 (CYP) 3A4 inhibitors or respiratory depressants, or could not safely discontinue these medications within 7 days or 5 half -lives (whichever is longer) prior to receiving study drug in the Qualification Phase and for the Duration of the study.
10. Subject was using an investigational drug or device or had used such within the 30 days (or 5 half-lives, whichever is longer) prior to first drug administration in the Qualification Phase.
11. Female subjects who were pregnant or lactating or who were planning to become pregnant within 14 days of last study drug administration.
12. Subject had a prior history of any significant adverse reactions (including rash) to benzodiazepines and/or flumazenil, or known allergies to midazolam and/or flumazenil, or formulation components.
13. Subject had unsuitable or difficult venous access or was unwilling or unable to undergo catheter insertion.
14. Subject was an employee of the sponsor or research site personnel directly affiliated with this study or their immediate family member defined as a spouse, parent, child, or sibling, whether biological or legally adopted.
15. A subject who, in the opinion of the investigator, was considered unsuitable or unlikely to comply with the study protocol for any reason (in each case, the investigator had to specify the reason).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 83 (Actual)
Dates: Start 2015-06-23 (Actual); Primary Completion 2015-10-06 (Actual); Study Completion 2015-10-06 (Actual)

PRIMARY OUTCOMES:
Drug Liking VAS maximum effect (Emax) | 2 to 480 minutes postdose
  Maximum effect (Emax) on the bipolar Drug Liking visual analogue scale (VAS)

SECONDARY OUTCOMES:
Drug Liking VAS Minimum effect [Emin] | 2 to 480 minutes postdose
  Minimum effect (Emin) on the bipolar Drug Liking visual analogue scale (VAS)
Overall Drug Liking VAS (Emax/Emin) | 240 to 480 minutes postdose
  Emax/Emin on the bipolar Drug Liking visual analogue scale (VAS)
Take Drug Again VAS (Emax) | 240 to 480 minutes postdose
  Maximum effect (Emax) on the unipolarTake Drug Again visual analogue scale (VAS)
Good Effects VAS (Emax and TA_AUE) | 2 to 480 minutes postdose
  Maximum effect (Emax) and TA_AUE on the unipolar Good Effects visual analogue scale (VAS)
Bad Effects VAS (Emax and TA_AUE) | 2 to 480 minutes postdose
  Maximum effect (Emax) and TA_AUE on the unipolar Bad Effects visual analogue scale (VAS)
Alertness/Drowsiness VAS (Emin and TA_AUE) | Predose to 480 minutes postdose
  Minimum effect (Emin) and TA_AUE on the bipolar Alertness/Drowsiness visual analogue scale (VAS)
Agitation/Relaxation VAS (Emin and TA_AUE) | Predose to 480 minutes postdose
  Minimum effect (Emin) and TA_AUE on the bipolar Agitation/Relaxation visual analogue scale (VAS)
Any Effects VAS (Emax and TA_AUE) | 2 to 480 minutes postdose
  Maximum effect (Emax) and TA_AUE on the unipolar Any Effects visual analogue scale (VAS)
Paired Associates Learning (PAL) total error score (Emax and TA_AUE) | Predose to 480 minutes postdose
  PAL test was conducted using the software CANTAB (Cambridge Cognition)

CONTACTS AND LOCATIONS:
Overall Officials: Shawn Searle, MD, Principal Investigator — PRA Health Sciences
Locations (1):
- PRA Health Sciences Early Development Services, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No